CLINICAL TRIAL: NCT04466397
Title: Repair of the Large Bone Defects Through 3D Printed Individualized Porous Implant: a New "Implant-bone" Interface Fusion Concept for Large Bone Defects Treatment
Brief Title: Repair of the Large Bone Defects Through 3D Printed Individualized Porous Implant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Liuzhongjun-1
Record Dates: First submitted 2020-06-28; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-06

CONDITIONS: Large Bone Defects
Keywords: large bone defects; 3D printed individualized porous implant; "implant-bone" interface fusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3D printed implants reconstruction group: The patients with large bone defects who treated by 3D printed individualized porous implants
  Interventions: Device: 3D printed individualized porous implants

INTERVENTIONS:
Device: 3D printed individualized porous implants — Use 3D printed individualized porous implants to reconstruct the large bone defects caused by tumor, infection or trauma.

SUMMARY:
The aim of this study was to investigate the simply use of three-dimensional (3D) printed individualized porous implants in the absence of autogenous/allogeneic bone graft or any osteoinductive agents to treat the large bone defects caused by varies of pathogenesis and systematically study its long-term therapeutic effect and osseointegration characteristics.

DETAILED DESCRIPTION:
A selection of fifty-eight patients with large bone defects caused by tumor, infection or trauma received the individualized porous implants treatment, and two typical cases were chosen for detailed study. Further, the large segmental femur defect model of sheep was utilized to study the osseointegration characteristics of the individualized porous implants in 1, 3, 6 months after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Large bone defects (>4cm) in spine, limb bone and hip joint caused by tumor, infection or other pathogenesis received the individualized porous implants treatment.Exclusion Criteria:
* Bone defects less than 4cm long.
* Bone defects treated by other methods ,such as ilizarov technique, masquelet technique or Ti mesh.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with bone tumor or bone infection who are diagnosed with large bone defects after receiving surgery in our Peking University Third Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Biomechanical stability | Immediate after the bone defect reconstruction.
  Evaluete the immediate and long-term biomechanical stability of the bone-implant complex after surgery by the following indicator: the loosening, subsidence, displacement of the implants from radiographic examination and The symptoms of the patient.
Biomechanical stability | 2 months after the bone defect reconstruction.
  Evaluete the immediate and long-term biomechanical stability of the bone-implant complex after surgery by the following indicator: the loosening, subsidence, displacement of the implants from radiographic examination and The symptoms of the patient.
Biomechanical stability | 5 months after the bone defect reconstruction.
  Evaluete the immediate and long-term biomechanical stability of the bone-implant complex after surgery by the following indicator: the loosening, subsidence, displacement of the implants from radiographic examination and The symptoms of the patient.
Biomechanical stability | 8 months after the bone defect reconstruction.
  Evaluete the immediate and long-term biomechanical stability of the bone-implant complex after surgery by the following indicator: the loosening, subsidence, displacement of the implants from radiographic examination and The symptoms of the patient.
Biomechanical stability | 14 months after the bone defect reconstruction.
  Evaluete the immediate and long-term biomechanical stability of the bone-implant complex after surgery by the following indicator: the loosening, subsidence, displacement of the implants from radiographic examination and The symptoms of the patient.
Biomechanical stability | 20 months after the bone defect reconstruction.
  Evaluete the immediate and long-term biomechanical stability of the bone-implant complex after surgery by the following indicator: the loosening, subsidence, displacement of the implants from radiographic examination and The symptoms of the patient.

SECONDARY OUTCOMES:
Osseointegration | Immediate after the bone defect reconstruction.
  Evaluate the osseointegration characteristics of the bone-implant complex by using CT scan to quantify the callus bridging at the outer surface of the implants or the bone growing into the porous implants.
Osseointegration | 2 months after the bone defect reconstruction.
  Evaluate the osseointegration characteristics of the bone-implant complex by using CT scan to quantify the callus bridging at the outer surface of the implants or the bone growing into the porous implants.
Osseointegration | 5 months after the bone defect reconstruction.
  Evaluate the osseointegration characteristics of the bone-implant complex by using CT scan to quantify the callus bridging at the outer surface of the implants or the bone growing into the porous implants.
Osseointegration | 8 months after the bone defect reconstruction.
  Evaluate the osseointegration characteristics of the bone-implant complex by using CT scan to quantify the callus bridging at the outer surface of the implants or the bone growing into the porous implants.
Osseointegration | 14 months after the bone defect reconstruction.
  Evaluate the osseointegration characteristics of the bone-implant complex by using CT scan to quantify the callus bridging at the outer surface of the implants or the bone growing into the porous implants.
Osseointegration | 20 months after the bone defect reconstruction.
  Evaluate the osseointegration characteristics of the bone-implant complex by using CT scan to quantify the callus bridging at the outer surface of the implants or the bone growing into the porous implants.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongjun Liu, Bachelor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No